CLINICAL TRIAL: NCT05741242
Title: A Phase 1b/2, Multi-center, Single Arm Study to Assess the Safety and Efficacy of Neoantigen Synthetic Long Peptide Vaccines in Patients With Local Or Metastatic Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jaime Leandro Foundation for Therapeutic Cancer Vaccines (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLF-200
Expanded Access: Available
Record Dates: First submitted 2021-08-16; First posted 2023-02-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Solid Tumor
Keywords: personalized neoantigen vaccine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Personalized Synthetic Long Peptide Vaccine (Experimental)
  Interventions: Biological: Personalized Synthetic Long Peptide Vaccine

INTERVENTIONS:
Biological: Personalized Synthetic Long Peptide Vaccine — Personalized Synthetic Long Peptide Vaccine

SUMMARY:
A Phase 1b/2, Multi-center, Single Arm Study to Assess the Safety and Efficacy of Neoantigen Synthetic Long Peptide Vaccines in Patients With Local Or Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a Simon-two stage multi-cohort study to assess the safety and efficacy of neoantigen synthetic long peptide vaccines in patients with local or metastatic solid tumors.

1. To assess the efficacy of NeoSLP vaccination by investigator assessment of Progression-Free Survival at 12 months (PFS12).
2. To assess efficacy of NeoSLP vaccination by assessment of Time to Treatment Failure (TTF).
3. To assess efficacy of NeoSLP vaccination by assessment of Overall Survival at 24 months (OS24).
4. To investigate the immunogenicity of NeoSLP vaccines by ELISpot assay. 5. To assess the safety and tolerability of NeoSLP vaccines.

ELIGIBILITY:
Patients must satisfy the following criteria to be enrolled in the protocol:

Main Inclusion Criterion:

Pancreatic

1. Patients who have local or metastatic pancreatic adenocarcinoma and have started first line therapy of Folfirinox (physician's choice for any concomitant therapies)
2. Patients who have undergone somatic tumor sequencing should consider FDA-approved pan-solid tumor therapies if they harbor an FDA-approved somatic alteration. For example, Entrectinib or Larotrectinib (if NTRK gene fusion- positive), Selpercatinib (if RET gene fusion-positive), Pembrolizumab (if MSI-H, dMMR, or TMB-H[≥10 mut/Mb]), and PARP inhibitors (BRCA mutations).

Glioblastoma

1. Patients who are within 6 months of diagnosis and have detectable disease as determined by investigator assessment at the start of vaccine administration.

Basket

1. Patients with local or metastatic malignancies, limited treatment options, and an estimated 5-year survival of less than 50% are eligible for enrollment in this cohort.

Other Inclusion Criteria:

1. >= 12 years of age.
2. ECOG performance status ≤ 2 or Karnofsky score of >=70.
3. Adequate organ function allowing favorable benefit to risk ratio per the treating physician
4. Systemic corticosteroid therapy is permitted provided dosing is no greater than 4 mg per day (dexamethasone or equivalent) on the day of vaccine administration.
5. Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. History of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty or known allergy to a component of the neoantigen synthetic long peptide vaccine.
2. Intercurrent illness requiring chronic use of medications that may interfere with rescue medications for treatment of vaccine-related anaphylaxis or attenuate immune response to vaccine treatment (immunosuppressive therapies).
3. Psychiatric illness or social situations that would limit compliance with study requirements.
4. History of pre-existing immunodeficiency disorder or autoimmune condition requiring immunosuppressive therapy that would preclude response to vaccine.
5. Females of childbearing potential may participate provided they agree to practice abstinence; and, if heterosexually active, agree to use at least 2 highly effective contraceptive methods throughout the study and for 3 months following the last dose of study drug; and have a negative serum pregnancy test.
6. Females of non-childbearing potential must be post-menopausal or have been surgically sterilized.
7. Male subjects with a female partner of childbearing potential must agree to practice abstinence or to use a physician-approved contraceptive method throughout the study and for 3 months following the last dose of study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of NeoSLP vaccination by investigator assessment of Progression-Free Survival at 12 months (PFS12). | Until progression or death, assessed up to 12 months post first vaccine administration.
  Progression-Free Survival at 12 months (PFS12) defined as time from first vaccine administration until disease progression by investigator assessment or death due to any cause.

SECONDARY OUTCOMES:
To assess efficacy of NeoSLP vaccination by assessment of Time to Treatment Failure (TTF). | Assessed up to 12 months post first vaccine administration
  Time to Treatment Failure (TTF) is defined as time from first vaccine administration to discontinuation of treatment due to any reason, including disease progression, treatment toxicity, and death.
To assess efficacy of NeoSLP vaccination by assessment of Overall Survival at 24 months (OS24). | Until death, assessed up to 24 months post first vaccine administration
  Overall Survival at 24 months (OS24) is the landmark of OS defined as the proportion of patients alive at 24 months.
To assess the safety and tolerability of NeoSLP vaccines. | Assessed up to 60 days from last vaccine administration
  Adverse Events (AEs) and Severe Adverse Events (SAEs)

OTHER OUTCOMES:
To investigate the immunogenicity of NeoSLP vaccines by ELISpot assay. | Assessed at baseline before first vaccine administration and day 50 post
  Immune monitoring is defined as the percentage of patients showing an immune response to the vaccine components.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Precision NextGen Oncology & Research Center, Beverly Hills, California
  - Quest Clinical Research, San Francisco, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - St. Louis Cancer Care, Bridgeton, Missouri
  - Anna Gattani MD PC, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided